CLINICAL TRIAL: NCT04750746
Title: Effects of Exer-gaming on Upper Extremity Function and Activities of Daily Living in Sub-acute Stroke Patient.
Brief Title: Exer-gaming on Upper Extremity Function and Activities of Daily Living in Sub-acute Stroke Patient.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/Lhr/20/2032 Yamna Mazhar
Record Dates: First submitted 2021-02-10; First posted 2021-02-11 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Stroke; Cardiovascular Stroke; Cerebrovascular Accident
MeSH Terms: conditions — Stroke; Myocardial Infarction | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Control group will get conventional treatment.
  Interventions: Other: Control group
- Experimental Group (Experimental): This group will get base line treatment with exer gaming.
  Interventions: Other: Experimental Group

INTERVENTIONS:
Other: Control group — Conventional Therapy Passive ROM and/or AROM exercises Muscle strengthening; Therapeutics stretching of the shoulder, the elbow, the wrist, and the fingers. Activities of daily living training, including eating, grooming, dressing, toileting, and transfer
  Arms: Control Group
Other: Experimental Group — Interventional therapy Xbox Kinect (Xbox 360, Microsoft,) For training, programs such as Boxing and Bowling in the Kinect sports pack and Rally Ball, 20,000 Leaks, and Space Pop in the Kinect adventure pack, all of which required the use of the upper extremities, will be selected
  Arms: Experimental Group

SUMMARY:
Stroke is one of the leading cause of death, in adult stroke causes permanent disability. Stoke impact the life of a person significantly including the quality of life of an individual and especially performing the task of daily activities independently. About 50% survival of stroke have daily life activity limitation which is affecting their quality of life. Among stroke patients, 69% experience functional motor disturbance in their upper extremity.

The aim of this study is to evaluate the effect of Exer-gaming by using the Xbox Kinect game system on upper extremity motor functions and the ability to perform ADLs in sub-acute stroke. Various treatment methods are used for the rehabilitation of stroke. This study will be a randomized controlled trial, used to compare the effectiveness of Exer gaming on upper extremity function and activities of daily living in sub-acute stroke patient. Subjects with Sub-acute stroke meeting the predetermined inclusion & exclusion criteria will be divided into two groups using simple random sampling technique. Pre assessment will be done using FMA & SIS measurements. Subjects in one group will be treated with Conventional therapy and exer gaming and the other will be treated with conventional therapy and activities training session. Each subject will be received a total 18 treatment sessions, with 3 treatment sessions per week for 6 weeks. Post treatment reading for FMA and SIS will be recorded after the end of treatment session. Recorded values will be analyzed for any change using SPSS.

ELIGIBILITY:
Inclusion Criteria:

* 1) First stroke 2) Patient of sub-acute stroke 3) Both gender 4) Between 45 to 65 years of age 6) Total score of 19 or greater on the Mini-Mental State Examination 7) No problems with auditory or visual functioning.

Exclusion Criteria:

* 1) Patient with global aphasia, and blindness, 2) Taking any prescribed drugs that could potentially affect physical function and balance (such as corticosteroids, antipsychotics or antidepressants) 3) Uncontrolled blood pressure (HTN) 4) Cardiac conditions 5) History of seizure 6) Any intervention other than conventional therapy 7) Refusal to use a video game.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-03-27 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
upper extremity function | 4 months
  The Fugl-Meyer Upper Extremity (FMUE) Scale1 is a widely used and highly recommended stroke-specific, performance-based measure of impairment. The FMUE Scale comprises 33 items, each scored on a scale of 0 to 2, where 0 = cannot perform, 1 = performs partially and 2 = performs fully.
Activities of daily living | 4months
  It was measured by stroke impact scale. The purpose of this questionnaire is to evaluate how stroke has impacted the health and life. On a scale of 0 to 100, with 100 representing full recovery and 0 representing no recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Iram Shafee, M.Phil, Principal Investigator — Riphah International University
Locations (1):
- Iram Shafee, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Henrique PPB, Colussi EL, De Marchi ACB. Effects of Exergame on Patients' Balance and Upper Limb Motor Function after Stroke: A Randomized Controlled Trial. J Stroke Cerebrovasc Dis. 2019 Aug;28(8):2351-2357. doi: 10.1016/j.jstrokecerebrovasdis.2019.05.031. Epub 2019 Jun 13. PMID 31204204
- [Background] Kim JH. Effects of a virtual reality video game exercise program on upper extremity function and daily living activities in stroke patients. J Phys Ther Sci. 2018 Dec;30(12):1408-1411. doi: 10.1589/jpts.30.1408. Epub 2018 Nov 21. PMID 30568325
- [Background] Trombetta M, Bazzanello Henrique PP, Brum MR, Colussi EL, De Marchi ACB, Rieder R. Motion Rehab AVE 3D: A VR-based exergame for post-stroke rehabilitation. Comput Methods Programs Biomed. 2017 Nov;151:15-20. doi: 10.1016/j.cmpb.2017.08.008. Epub 2017 Aug 12. PMID 28946996
- [Background] Nguyen AV, Ong YA, Luo CX, Thuraisingam T, Rubino M, Levin MF, Kaizer F, Archambault PS. Virtual reality exergaming as adjunctive therapy in a sub-acute stroke rehabilitation setting: facilitators and barriers. Disabil Rehabil Assist Technol. 2019 May;14(4):317-324. doi: 10.1080/17483107.2018.1447608. Epub 2018 Mar 12. PMID 29529895
- [Background] Sin H, Lee G. Additional virtual reality training using Xbox Kinect in stroke survivors with hemiplegia. Am J Phys Med Rehabil. 2013 Oct;92(10):871-80. doi: 10.1097/PHM.0b013e3182a38e40. PMID 24051993
- [Background] Ahmad MA, Singh DKA, Mohd Nordin NA, Hooi Nee K, Ibrahim N. Virtual Reality Games as an Adjunct in Improving Upper Limb Function and General Health among Stroke Survivors. Int J Environ Res Public Health. 2019 Dec 16;16(24):5144. doi: 10.3390/ijerph16245144. PMID 31888293
- [Background] Warland A, Paraskevopoulos I, Tsekleves E, Ryan J, Nowicky A, Griscti J, Levings H, Kilbride C. The feasibility, acceptability and preliminary efficacy of a low-cost, virtual-reality based, upper-limb stroke rehabilitation device: a mixed methods study. Disabil Rehabil. 2019 Sep;41(18):2119-2134. doi: 10.1080/09638288.2018.1459881. Epub 2018 Apr 12. PMID 29644897